CLINICAL TRIAL: NCT04209751
Title: Descriptive Study of Pathogens Involved in Summer Diarrhea in Children Leading to Pediatric Emergency Room Visits
Brief Title: Descriptive Study of Pathogens Involved in Summer Diarrhea in Children Leading to Pediatric Emergency Room Visits (PE-DIA)
Acronym: PE-DIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Society ELITECH (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 VERDAN; 2019-A02341-56 (Other: ANSM)
Record Dates: First submitted 2019-11-28; First posted 2019-12-24 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-09

CONDITIONS: Diarrhea, Infantile
Keywords: Microbiologic diagnosis; summer diarrhea; pediatric population
MeSH Terms: conditions — Diarrhea, Infantile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with summer diarrhea: Children aged 0 to 16 years with diarrhea
  Interventions: Diagnostic Test: Stool removal

INTERVENTIONS:
Diagnostic Test: Stool removal — Stool removal; freezing an aliquot at -20 ° C and performing a direct examination. DNA extraction and serial PCR (Polymerase chain reaction).

SUMMARY:
Acute diarrhea in children is a public health problem. It is estimated that children under 3 years are subject to 1 or 2 episodes of diarrhea per year in Europe. These diarrheal episodes are frequent, expensive and responsible for many consultations and hospitalizations in developed countries. The origin of diarrhea in children is viral in about 70% of cases. The diagnosis of a viral infection is often considered without microbiological evidence. However, microbiological evidence is recommended for certain categories of patients.

The involvement of bacteria or parasites in the child's diarrhea does not seem negligible.

The main objective of this study is to estimate the prevalence of infectious diarrhea among summer diarrhea in children leading to pediatric emergency room visits.

Secondarily, we will describe the pathogens responsible for childhood diarrhea during the summer period, describe common factors that can serve as guidance on the etiology of diarrhea, and describe common factors that can be used as tools. preventive to the transmission of these pathogens.

DETAILED DESCRIPTION:
After obtaining consent from the holders of parental authority, a stool collection will be requested from all pediatric emergency patients presenting as a reason for "diarrhea" consultations between June 1 and September 30, 2020. It will be given by the nurse organizing the reception, a medical information questionnaire and a stool collection container for those accompanying a child with diarrhea.

If the child presents stool during the waiting period or during the medical consultation, these will be collected and sent to the medical biology laboratory of the University Hospital for a broad analysis (virological, bacteriological and parasitological).

The doctor in charge of the patient will complete a pre-established clinical information sheet.

In the laboratory, the stool will be taken care of and a DNA extract will be made and preserved. The search for pathogens will be carried out by molecular biology, by series, non-prospectively. The results will only be transmitted at a distance and will not be communicated to families.

Therapeutic management of children included in the study will be identical to the usual practice. Microbiological analysis will not delay, prolong or disrupt the treatment of the acute episod of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 0 to 16 years with diarrhea
* pediatric emergency at the University Hospital of Clermont-Ferrand consultation
* between june and september 2020

Exclusion Criteria:

* consent not felt by the child or the person with parental authority
* no stool removal

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from 0 to 16 years with diarrhea
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of infectious diarrhea in children who consult pediatric emergencies in summerdiarrhea leading to pediatric emergency room visits | Day 0
  percentage of positive stool tests (PCR (polymerase chain reaction) and direct microscopic examination)Stool sent instantly to the laboratory. Microbological research : PCR and direct microscopic examination.

SECONDARY OUTCOMES:
Describe pathogens found in stool | Day 0
  Identification of pathogens by PCR and direct microscopic examination.
Describe common factors that can serve as preventive tools for the transmission of these pathogens. | Day 0
  prospective analyzes of data collected from parental authority using a questionnaire
Describe common factors that can be used as guidance on the etiology of diarrhea | Day 0
  prospective analyzes of the data collected from the parental authority and causal link with a specific germ

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Verdan, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France